CLINICAL TRIAL: NCT07145385
Title: Prevalence of Alpha-1 Antitrypsin Deficiency in a Cohort of Hepatocellular Carcinoma on Non-Cirrhotic Liver Without Identified Etiologies
Brief Title: Prevalence of Alpha-1 Antitrypsin Deficiency in Non-Cirrhotic Liver Cancer
Acronym: CHAMAD
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2024/43
Record Dates: First submitted 2025-06-27; First posted 2025-08-28 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Retrospective Cohort of Patients Diagnosed With HCC on Non-Cirrhotic Liver
Keywords: Prevalence; Alpha-1 Antitrypsin Deficiency; HCC on Non-Cirrhotic Liver; Retrospective Cohort
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients Diagnosed with HCC on Non-Cirrhotic Liver: Patients Diagnosed with HCC on Non-Cirrhotic Liver
  Interventions: Other: multiplex digital PCR

INTERVENTIONS:
Other: multiplex digital PCR — multiplex digital PCR

SUMMARY:
Patients with Alpha-1 Antitrypsin Deficiency (AATD), a rare genetic disease, have a 20- to 50-fold higher risk of developing primary liver cancer (PLC), such as hepatocellular carcinoma (HCC), in both cirrhotic and non-cirrhotic livers, highlighting AATD as a potential oncogenic factor. Therefore, our aim is to evaluate the association between AATD and HCC in patients with a non-cirrhotic liver and no known predisposition

DETAILED DESCRIPTION:
The two most common pathogenic AATD variants, PiS and PiZ, will be identified using the multiplex digital PCR (dPCR) system in a French cohort of 71 patients who developed HCC in a non-cirrhotic liver without known risk factors for HCC

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (≥18 years of age).
2. Histopathologically confirmed diagnosis of hepatocellular carcinoma (HCC).
3. Normal liver or chronic liver disease with minimal to moderate fibrosis in non-tumoral tissue.
4. Signed informed consent obtained prior to participation.
5. No other known etiology or risk factors for liver disease, including:

   * Alcohol-related liver disease
   * Metabolic-associated steatohepatitis (MASH)
   * Viral hepatitis infections
   * Hemochromatosis

Exclusion Criteria:

1. Minor patients (<18 years of age).
2. HCC diagnosis not established according to standard histopathological criteria.
3. Liver with chronic liver disease showing advanced fibrosis in non-tumoral tissue.
4. No signed informed consent prior to participation.
5. Presence of other identified etiologies or known risk factors for liver disease, including:

   * Alcohol-related liver disease
   * Metabolic-associated steatohepatitis (MASH)
   * Viral hepatitis infections
   * Hemochromatosi

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients Diagnosed with HCC on non-cirrhotic liver
Sampling Method: Non-Probability Sample
Enrollment: 71 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Alpha-1 Antitrypsin Deficiency | 1 year
  Prevalence of Alpha-1 Antitrypsin Deficiency in a Retrospective Cohort of Patients Diagnosed with HCC on Non-Cirrhotic Liver up to 1 year

SECONDARY OUTCOMES:
Correlation of clinico-biological parameters-including survival (years), sex, BMI, fibrosis stage, mode of diagnosis, number of tumors, tumor size (mm), metastasis, recurrence, and Edmondson score-according to AAT genotype | 1 year
  Correlation of clinico-biological parameters-including survival (years), sex, BMI, fibrosis stage, mode of diagnosis, number of tumors, tumor size (mm), metastasis, recurrence, and Edmondson score-according to AAT genotype. up to 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Bordeaux, Bordeaux, France